CLINICAL TRIAL: NCT01591226
Title: Effects of Caffeine and Sodium Citrate Ingestion in 1500m Wheelchair Racing Athletes
Brief Title: Caffeine and Sodium Citrate Ingestion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012-02
Record Dates: First submitted 2012-04-03; First posted 2012-05-03 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Dietary Supplements; Heart Rate/Drug Effects; Lactic Acid/Metabolism; Physical Education and Training/Methods; Wheelchairs
Keywords: caffeine; sodium citrate; exercise performance; wheelchair athletes; 1500m
MeSH Terms: interventions — Caffeine; Sodium Citrate; Mannitol; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Caffeine (Active Comparator): 6mg per kg bodyweight ingested 60min before test
  Interventions: Dietary Supplement: Caffeine; Dietary Supplement: Sodium Chloride
- Placebo (Placebo Comparator): Sodium chloride and mannitol as placebo are ingested by the athlete
  Interventions: Dietary Supplement: Mannitol; Dietary Supplement: Sodium Chloride
- Sodium Citrate (Active Comparator): sodium citrate diluted in 7dl water, ingestion 120 to 90min prior test
  Interventions: Dietary Supplement: Sodium Citrate; Dietary Supplement: Mannitol
- Caffeine and Sodium Citrate (Active Comparator): sodium citrate 120-90min prior test capsules:60min prior test
  Interventions: Dietary Supplement: Caffeine; Dietary Supplement: Sodium Citrate

INTERVENTIONS:
Dietary Supplement: Caffeine — gelatine capsule 6mg/kg bodyweight 60min prior test
  Arms: Caffeine; Caffeine and Sodium Citrate
Dietary Supplement: Sodium Citrate — 0.5g/kg bodyweight diluted in 7dl water ingested 120-90min prior test
  Arms: Caffeine and Sodium Citrate; Sodium Citrate
Dietary Supplement: Mannitol — gelatine capsule filled with mannitol (100mg per capsule) ingested 60min prior test
  Arms: Placebo; Sodium Citrate
Dietary Supplement: Sodium Chloride — sodium chloride diluted in 7dl water 0.045g/kg bodyweight 120-90min prior test
  Arms: Caffeine; Placebo

SUMMARY:
A positive ergogenic effect of sodium citrate and caffeine ingestion in a short-term, high-intensity exercise task was shown by several studies. These studies were conducted with healthy, able-bodied subjects.

The aim of the study is to investigate whether caffeine or sodium citrate ingestion could enhance performance in spinal cord injured wheelchair athletes. It is a double blind, placebo controlled and randomized study.

DETAILED DESCRIPTION:
The athletes have to complete four 1500m tests on a training roller. Before each treatment they get different supplementations. Once they get sodium citrate and a placebo, once caffeine and a placebo, once sodium citrate and caffeine and for the fourth treatment they get twice a placebo. Two hours after starting with the supplementation they have to complete the 1500m as fast as possible. Time to complete 1500m, blood pH, plasma bicarbonate, sodium concentration, heart rate, oxygen consumption, blood lactate concentration and rate of perceived exertion (RPE) were measured.

ELIGIBILITY:
Inclusion Criteria:

* wheelchair athletes
* national team
* category T53 and T54

Exclusion Criteria:

* medicated
* pregnant (for women)
* cardiovascular and respiratory diseases

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2012-02; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Time | 3 weeks
  Time to complete 1500m

SECONDARY OUTCOMES:
Heart Rate | during study phase of 3 week (4 tests)
  Heart Rate measured from 2min before the test until 5min after the 1500m-test.
Lactate Concentration | during the 3 weeks study phase
  1min before starting the warm up, 15s after the end of the warm up, 15s after completing the test, 2min/4min/6min/8min/10min after the test
blood pH, sodium concentration and plasma bicarbonate | during the 3 weeks of study phase
  1min before starting with the ingestion of the fluid, immediately before starting the warm up, just immediately before starting the 1500m test.
Oxygen Consumption | during 3 weeks of study phase
  oxygen consumption (VO2(ml/min/kg), VCO2(ml/min), RER (VCO2/VO2)) starting of the measurement is 2min before the start of the 1500m and ends 2min after having completed the 1500m
rating of gastrointestinal stress | during the 3 weeks of study phase
  1min before starting to drink the fluid, 2min before starting with the warm up, 2min before the test and 2min after having completed the 1500m
Rating of Perceived Exertion (RPE) | during the 3 weeks of study phase
  15s after the end of the warm up, 15s after having completed the 1500m

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Perret, Dr. sc. nat., Principal Investigator — Swiss Paraplegic Research, Nottwil
Locations (1):
- Swiss Paraplegic Centre, Nottwil, Canton of Lucerne, Switzerland